CLINICAL TRIAL: NCT04123236
Title: Investigation of the Relationship of Orthodontic Malocclusions With Temporomandibular Joint Disorders by Helkimo's Indices and Oral Health Impact Profile-14
Brief Title: The Relationship of Orthodontic Malocclusions With Temporomandibular Joint Disorders
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Aysegul Gulec, Principal investigator, University of Gaziantep
Other Study IDs: 81
Record Dates: First submitted 2019-10-02; First posted 2019-10-10 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-12

CONDITIONS: Temporomandibular Joint Disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — lobo protein, Drosophila

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Oral Health Impact Profile: To evaluate the Oral Health-related Quality of Life, Turkish version of Oral Health Impact Profile-14 was used. Responses were made on a scale 0 (never), 1(hardly ever), 2 (occasionally), 3 (fairly often),and 4 (very often).Oral Health-related Quality of Life impairment was characterized by the Oral Health Impact Profile-14 summary score (the sum of all 14 items, potential range 0-56). Higher Oral Health Impact Profile-14 scores mean worse Oral Health-related Quality of Life and vice versa.
  Interventions: Other: Age 0-18; Other: Age 18-26; Other: Girls; Other: Boys
- Helkimo's anamnestic dysfunction index: As a method based on patient feedback for the determination of the degree of temporomandibular disorders, anamnestic index was used. For this purpose eight questions were asked to the patients that includes answers as 'yes' or 'no'. (Table 2) The analyses of the questionnaire was done according to anamnestic scale as 0: no symptoms; I: mild symptoms (sensation of the jaw fatigue, jaw stiffness, and temporomandibular joint sounds as clicking or crepitus) and II:severe symptoms (included one or more of the following: Difficulty in the mouth opening, jaw locking, mandible dislocation and its painful movement and painful temporomandibular joint region and/or masticatory muscles)
  Interventions: Other: Age 0-18; Other: Age 18-26; Other: Girls; Other: Boys
- Visual analog scale (VAS) for facial pain:: Facial pain was measured by asking the patients if they had had any pain during last 12 months and made them mark the intensity of the pain on a visual analog scale which had the anchor points at the left (no pain) and right (worse pain) ends of a 10 cm horizontal line. The analyses of the facial pain was done as fallowing: if the patient marked no facial pain the Visual analog scale value was accepted as 0 and if the patient marked any level of facial pain Visual analog scale value was accepted as 1.
  Interventions: Other: Age 0-18; Other: Age 18-26; Other: Girls; Other: Boys
- Helkimo's clinical dysfunction index (DI):: Maximum opening of mandible, deviation during opening, dysfunction of temporomandibular joint, pain in the temporomandibular joint and pain in the masticatory muscles was evaluated
  Interventions: Other: Age 0-18; Other: Age 18-26; Other: Girls; Other: Boys

INTERVENTIONS:
Other: Age 0-18 — Patients under 18 years of age
Other: Age 18-26 — Patients over18 years of age
Other: Girls — Girls
Other: Boys — Boys

SUMMARY:
The patients who applied to the hospital for orthodontic treatment were asked various questions to evaluate their oral health related quality of life, malocclusions and self reported temporomandibular joint problems.

DETAILED DESCRIPTION:
The patients who applied to the hospital for orthodontic treatment were asked various questions to evaluate their oral health related quality of life, malocclusions and self reported temporomandibular joint problems. For this purposes Oral Health Impact Profile-14, and Helkimo's indexes were used.The relationship between these results were investigated.

ELIGIBILITY:
Inclusion Criteria:

* wish to receive orthodontic treatment in our clinic.

Exclusion Criteria:

* The absence of willingness for the temporomandibular joint and clinical examination or answering the survey questions.

Ages: 12 Years to 27 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients wish to receive orthodontic treatment in our clinic.
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2019-07-20 (Actual); Study Completion 2020-10-20 (Estimated)

PRIMARY OUTCOMES:
Oral Health Impact Profile | through study completion, an average of 2 months. The scale ranged from 0-5. All data will be summed at the end of the study. Higher values means worse quality of life standard
  Oral Health Impact Profile relations between patients under 18 and over 18 and between girls and boys
Helkimo's anamnestic dysfunction index | through study completion, an average of 2 months. The scale ranged from 0-3. Higher scale means worse quality of life standards
  Helkimo's anamnestic dysfunction index relations between patients under 18 and over 18 and between girls and boys
Helkimo's clinical dysfunction index | through study completion, an average of 2 months. The scale ranged from 0-3. Higher scale means worse quality of life standards
  Helkimo's clinical dysfunction index relations between patients under 18 and over 18 and between girls and boys
Visual analog scale | through study completion, an average of 2 months.
  Visual analog scale relations between patients under 18 and over 18 and between girls and boys. The scale ranged from 0-1. If the patient marked no facial pain the visual analog scale value was accepted as 0, if the patient marked any level of facial pain visual analog scale value was accepted as 1.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Goymen, PhD, Study Chair — University of Gaziantep; Yeşim Kaya, Study Chair — Yuzuncu Yil University
Locations (1):
- Gaziantep University, Gaziantep, Şehitkamil, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No